CLINICAL TRIAL: NCT02599467
Title: Evoked EMG Muscle Activity at Performing ULTN 1 in Breast Cancer Patients
Brief Title: EMG at Performing ULTN 1 in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, IRENE DE LA ROSA DÍAZ, PhD student, University of Alcala
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IDLR1985
Record Dates: First submitted 2015-09-15; First posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Physiotherapy
Keywords: Nerve Pain; Electromyography; Median Nerve; Breast Neoplasms
MeSH Terms: conditions — Neuralgia; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- case group 1: ALND (Experimental): Inclusion criteria: unilateral breast cancer surgery with Axillary lymph node dissection (ALND) during the last year and a half. Exclusion criteria: bilateral breast cancer, ipsilateral shoulder pathology, neuropathy.
  Procedure: ULNT 1 and EMG recording.
  Interventions: Other: ULNT 1 and EMG recording
- case group 2: SLNB (Experimental): Inclusion criteria: unilateral breast cancer surgery with Sentinel Lymph Node Biopsy (SLNB) during the last year and a half. Exclusion criteria: bilateral breast cancer, ipsilateral shoulder pathology, neuropathy.
  Procedure: ULNT 1 and EMG recording
  Interventions: Other: ULNT 1 and EMG recording
- control group (Active Comparator): Matched by age and dominant arm to each case. Exclusion criteria: current painful conditions involving their neck or dominant upper-extremity, and chronic pain conditions or use of pain relievers.
  Procedure: ULNT 1 and EMG recording.
  Interventions: Other: ULNT 1 and EMG recording

INTERVENTIONS:
Other: ULNT 1 and EMG recording — While the ULNT 1 was performing, EMG muscle activity form biceps brachii and triceps brachii were recorded. The maneuver was stopped to measure abduction, external rotation and elbow flexion range of motion (ROM) with a goniometer. Three measurements were performed: measure 1) when the first sense of tightness perceived by the subject appeared; measure 2) when evoked muscle activity increased on EMG record; measure 3) when sense of final resistance perceived by the investigator appeared. Considering the increase of symptoms with contralateral or decrease of symptoms with ipsilateral cervical side bending as mandatory positivity criterion.

SUMMARY:
Upper limb neural mechanosensitivity is a painful disturbance that breast cancer patients often undergo following axillary surgery. It is assessed by the upper limb neurodynamic test for the median nerve, called upper limb neurodynamic test 1 (ULNT1). Design: A matched case-control observational study. Objective: to check the increased upper limb mechanosensitivity by shoulder range of motion (ROM) during ULNT1 and to determine, for the first time, the evoked electromyographic (EMG) muscle activity. Participants: 62 cases who underwent breast cancer surgery and 64 matched control women. Setting: Torrejon Hospital, Physical Therapy Department, Madrid (Spain). Intervention: To record EMG muscle activity during ULNT1 performance and to measure shoulder ROM. Key outcomes: mechanosensitivity, breast cancer, pain, EMG, shoulder ROM, median nerve.

DETAILED DESCRIPTION:
Upper limb neural mechanosensitivity is a painful disturbance that breast cancer patients often undergo following axillary surgery. It is assessed by the upper limb neurodynamic test for the median nerve, called upper limb neurodynamic test 1 (ULNT1).A neural provocation test is a sequence of movements designed to assess the mechanics and physiology of part of the nervous system by elongating the length of the nerve bedding and by increasing the pressure in and around the peripheral nerve .The most reliable test to assess the upper limb neural mechanosensitivity is the neural provocation test for the median nerve, called upper limb neurodynamic test 1 (ULNT1). This test consists of depressing shoulder girdle in a neutral position, shoulder abduction and lateral rotation, elbow extension, forearm supination and wrist extension. Cervical contralateral lateral flexion may be included to further increase the loading of the brachial plexus and, as a sensitizing maneuver, to differentiate structurally between neural and non-neural involvement. The ULNT1 is considered as positive when symptoms are reproduced on affected upper limb, or side-to-side differences in ROM, or symptoms modified by lateral neck side-bending. Likewise, It is also necessary to assess the EMG activity of the involved muscles to verify the early and increased protective muscle response suggested throughout the neural strain performance.

It is also necessary to assess the EMG activity of the involved muscles to verify the early and increased protective muscle response suggested throughout the neural strain performance. Design: A matched case-control observational study. Objective: to check the increased upper limb mechanosensitivity by shoulder ROM during ULNT1 and to determine, for the first time, the evoked EMG muscle activity. Participants: 62 cases who underwent breast cancer surgery and 64 matched control women. Setting: Torrejon Hospital, Physical Therapy Department, Madrid (Spain). Intervention: To record EMG muscle activity during ULNT1 performance and to measure shoulder ROM. Key outcomes: mechanosensitivity, breast cancer, pain, EMG, shoulder ROM, median nerve.

ELIGIBILITY:
Inclusion Criteria:

* No undergo breast cancer.
* To be the age and the sema dominant arm than one of the cases.

Exclusion Criteria:

* Current painful conditions involving their neck or dominant upper-extremity.
* Chronic pain conditions (i.e. Fibromyalgia).
* Current use of pain relievers.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Increased evoked EMG muscle activity | 5 min
  Intensity of the evoked muscle activity from biceps brachii and triceps brachii muscles by EMG recording

SECONDARY OUTCOMES:
Upper limb range of motion restrictions | 15 min
  degrees of range of motion of three movements: shoulder abduction, shoulder external rotation and elbow flexion.

CONTACTS AND LOCATIONS:
Overall Officials: María Torres-Lacomba, Doctor, Study Director — Universidad Alcala